CLINICAL TRIAL: NCT06955910
Title: Assessing Financial Toxicity Using the PROFFIT Questionnaire in Patients Treated With Mini-invasive Approach for Urological Malignancies. UROFIT Study.
Brief Title: Assessing Financial Toxicity Using the PROFFIT Questionnaire in Patients Treated With Mini-invasive Approach for Urological Malignancies.
Status: Recruiting | Type: Observational
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IOV-UC-01-2025-UROFIT
Record Dates: First submitted 2025-04-16; First posted 2025-05-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Bladder Cancer; Kidney Cancer
Keywords: financial toxicity; PROFFIT questionnaire; robotic surgery; urological tumors; Prostate Cancer; Bladder Cancer; Kidney Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Financial Stress | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PROFFIT and EORTC QLQ-C30 questionnaires
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Anamnestic and socio-demographic information will be collected through a generic self-designed questionnaire including the following data: age, sex, residence (within or outside the Veneto region), marital status (married, divorced, cohabiting, single, widowed), employment status (employed, unemployed, retired), presence of dependents (yes/no), level of education (defined as primary, middle or high school, university degree), concomitant pathologies.
  Additional data on the oncological history are also reported: histology and staging of the disease, presence or absence of metastatic disease, additional treatments before or after surgery (e.g. neoadjuvant treatments, adjuvant treatments, radiotherapy).

SUMMARY:
Patients previously treated with robotic surgery for urological cancers such as prostate, bladder and kidney cancer will be enrolled, in particular patients operated in the last twelve months will be included after signing the informed consent.

Within 12 months after mini-invasive procedure, subjects are identified, contacted by phone/email, or invited to attend during the regular scheduled follow-up visit. If this is not possible, patients will be asked to schedule a special interview to assess possible participation in the study. During follow-up or unscheduled visit, the subsequent information will be collected through a questionnaire that contains several socio-demographic and anamnestic questions.

During subsequent visit, PROFFIT and EORTC QLQ-C30 questionnaires will be administered to patients. Post-operative complications are reported using the Clavien-Dindo classification.

Anamnestic and socio-demographic information will be collected through a generic self-designed questionnaire including the following data: age, sex, residence (within or outside the Veneto region), marital status (married, divorced, cohabiting, single, widowed), employment status (employed, unemployed, retired), presence of dependents (yes/no), level of education (defined as primary, middle or high school, university degree), concomitant pathologies.

Additional data on the oncological history are also reported: histology and staging of the disease, presence or absence of metastatic disease, additional treatments before or after surgery (e.g. neoadjuvant treatments, adjuvant treatments, radiotherapy).

DETAILED DESCRIPTION:
The rationale behind the design of this study is to define a snapshot of the impact of robotic surgery performed in uro-oncology patients on financial toxicity assessed through PROFFIT questionnaire. The design of a cross-sectional study allows to define whether minimally invasive surgical treatment can impact financial toxicity in a cohort of patients previously treated with minimally invasive surgery (which may differ for additional treatments received, ease of access to medical care secondary to place of residence/domicile, level of education, employment and family status).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age;
* ECOG PS 0-1
* Diagnosis of urological neoplasm (prostate, bladder and kidney cancer) treated with robotic surgery (robot-assisted prostatectomy, robot-assisted radical cystectomy, robot-assisted radical or partial nephrectomy) in the last twelve months;
* Subjects willing to sign informed consent.

Exclusion Criteria:

* Patients unable to fill out questionnaires (e.g., severe mental illness or cognitive dysfunction);
* Patients suffering from concomitant malignancies in other sites and in active treatment;
* Patients with a history of cancer not currently on active treatment may be enrolled.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: It is planned that the study will enroll about 120 Patients.
  In particular, patients with urological tumors who underwent minimally invasive surgery, using a robotic approach, in the last twelve months, will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Objective and end point | Through study completion, an average of 1 year
  Assess financial toxicity using the PROFFIT questionnaire in patients treated with robotic surgery for urological tumors. The PROFFIT questionnaire comprises the financial toxicity score (composed of the first 7 items) plus 9 other individual items indicating the possible determinants of financial difficulties. These items cover three main areas, such as medical expenses (items 8 to 11), transportation (items 12 and 13), and support for medical/health personnel (items 14 to 16).

SECONDARY OUTCOMES:
Secondary Objective and end point | Through study completion, an average of 1 year
  Evaluate factors associated to increased financial toxicity. Evaluation of the correlation between subjects' demographic characteristics and Financial Toxicity score (first 7 items)
Secondary Objective and end point | Through study completion, an average of 1 year
  Explore the correlation between financial toxicity and the impact on patients' quality of life. The EORTC QLQ-C30 questionnaire will be used to assess the patient's quality of life. This questionnaire has solid psychometric properties deriving from its use in several international clinical trials on cancer. Item Q28 and items Q29-30, the latter expressed according to "health status/quality of life scale" (HR-QoL), will be correlated with the FT score to assess the impact of financial toxicity on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto, Padua, Italy/Padova, Italy

IPD SHARING:
Plan to Share IPD: Undecided